CLINICAL TRIAL: NCT03034226
Title: A Comparison Between Counter Regulatory Responses in Type 1 Diabetic Patients Versus Healthy Control Subjects With and Without Antecedent Hypoglycemia
Brief Title: Comparison Between Hypoglycemic Counter Regulatory Responses in Type 1 Diabetics vs Control Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Project 1-10-72-304-16
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2018-03

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: Hypoglycemia-Associated Autonomic Failure (HAAF)
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Intervention Model Description: 9 diabetic subjects and 9 healthy control subjects will be randomized to undergo either first day 1 + day 2 (two consecutive episode of hypoglycemia) or first day 3 + day 4 (one episode of hypoglycemia).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single episode of hypoglycemia (Active Comparator): Day 1: Hyperinsulinemic hypoglycemic clamp 30 min Day 2: Hyperinsulinemic euglycemic clamp and hyperinsulinemic hypoglycemic clamp 7 hours
  Interventions: Other: Glucose clamp technique
- Two episodes of hypoglycemia (Active Comparator): Day 3: No intervention (normal blood glucose) Day 4: Hyperinsulinemic euglycemic clamp and hyperinsulinemic hypoglycemic clamp 7 hours
  Interventions: Other: Glucose clamp technique

INTERVENTIONS:
Other: Glucose clamp technique — Hyperinsulinemic euglycemic and hyperinsulinemic hypoglycemic clamp procedure with infusion of insulin and glucose

SUMMARY:
This study compares the hypoglycemic counter regulatory response in type 1 diabetics and in healthy control subjects with and without antecedent hypoglycemia

DETAILED DESCRIPTION:
Iatrogenic hypoglycemia is one of the main limiting factors for optimal glycemic management of diabetes. It causes recurrent morbidity in most people with type 1 diabetes and in many patients with type 2 diabetes and can be fatal. Episodes of hypoglycemia impair physiologically protective mechanism in subsequent episodes of hypoglycemia. This phenomenon is known as hypoglycemia-associated autonomic failure (HAAF), the clinical syndromes of defective glucose counter regulation and hypoglycemia unawareness.

ELIGIBILITY:
Type 1 diabetics

Inclusion Criteria:

* More than 5 years of disease duration
* HbA1c 42-86 mmol/L
* No known HAAF
* BMI 22-28
* Written consent

Exclusion Criteria:

* Other disease than diabetes f.x epilepsy, ischemic heart disease or heart rhythm disturbance
* Medication f.x beta-blockade, steroids, psychotropics
* Smoking
* Drug abuse

Control subjects

Inclusion Criteria:

* BMI 22-28
* Written consent

Exclusion Criteria:

* Diseases f.x diabetes, epilepsy, ischemic heart disease or heart rhythm disturbance
* Medication f.x beta-blockade, steroids, psychotropics
* Smoking
* Drug abuse

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Day 2 and day 4 (T=60 minutes - T=240 minutes)
  Insulin sensitivity before, during hypoglycemia and after recovery from hypoglycemia on day 2 (one episode of hypoglycemia) compared with day 4 (two consecutive episodes of hypoglycemia). Insulin sensitivity is measured as M-value derived from the Glucose Infusion Rate (GIR) during a hyperinsulinemic euglycemic clamp / hyperinsulinemic hypoglycemic clamp

SECONDARY OUTCOMES:
Hormonal counter regulatory response to hypoglycemia | Day 2 and day 4 (T=0 minutes, T=30, T=40, T=50, T=120, T=130, T=140, T160, T=170, T=180, T=210, T=220, T=230, T=390, T=400 and T=410
  Hormonal counter regulatory response (epinephrine, norepinephrine, glucagon, cortisol, ghrelin etc.) measured regularly before, during and after a hyperinsulinemic euglycemic clamp / hyperinsulinemic hypoglycemic clamp
Symptoms during hypoglycemia | Day 2 and day 4 (T=0 minutes - T=420 minutes)
  Using the Edinburgh Hypoglycemia Scale (symptom scale) we will interview the subjects regularly before, during and after a hyperinsulinemic euglycemic clamp / hyperinsulinemic hypoglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Mads Bisgaard Bengtsen, MD, phd student, Principal Investigator — Department of Endocrinology and Internal Medicine
Locations (1):
- Department of Clinical Medicine, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bengtsen MB, Stoy J, Rittig NF, Voss TS, Magnusson NE, Svart MV, Jessen N, Moller N. A Human Randomized Controlled Trial Comparing Metabolic Responses to Single and Repeated Hypoglycemia in Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa645. doi: 10.1210/clinem/dgaa645. PMID 32927476